CLINICAL TRIAL: NCT02955823
Title: A Combination of Lenalidomide and Rituximab as Front Line Therapy for the Treatment of Elderly Frail Patients Evaluated in CGA With Diffuse Large B-cells Non-Hodgkin Lymphoma. A Phase II Study of the Fondazione Italiana Linfomi (FIL)
Brief Title: A Phase II Study of the FIL on Elderly Frail Patients With DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_ReRi
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Diffuse Large B-cells Non-Hodgkin Lymphoma
Keywords: B cell Lymphoma; non-Hodgkin Lymphoma; Elderly patients
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 arm for all patient: Ritux-Dexame-Lena (Experimental): Rituximab-Dexamethasone-Lenalidomide
  Interventions: Drug: Rituximab-Dexamethasone-Lenalidomide

INTERVENTIONS:
Drug: Rituximab-Dexamethasone-Lenalidomide — 1. st CYCLE: Rituximab 375 mg/m2 i.v. on days 1,8,15; Dexamethasone 5 mg p.o. on days 1,8,15,22; Lenalidomide 15 mg/day p.o. day 2-22
  2. nd-4th CYCLE: Rituximab 375 mg/m2 i.v. on day 1; Lenalidomide 20 mg/day p.o. from day 2 to day 22 At the end of 4th CYCLE disease restaging: - if ≥ PR continues with the 5th and 6th cycle: Rituximab 375 mg/m2 i.v. on day 1, Lenalidomide 20 mg /day p.o. day 2-22
     * if <PR stops the treatment, only follow-up At the end of the 6th CYCLE disease restaging: - if ≥ PR continues with beyond the 6th cycle with Lenalidomide 10mg dd1-21q28 until cycle 12th
     * if <PR stops the treatment, only follow-up Then, accordingly response rate after the sixth cycle assessment(≥ PR) lenalidomide will be continued at 10 mg dd1-21q28 until 12th cycle or unacceptable toxicity.

SUMMARY:
A phase II study to evaluate the combination of Lenalidomide and Rituximab as front line therapy for the treatment of elderly frail patients evaluated in CGA with Diffuse Large B-cells non-Hodgkin Lymphoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm, phase II trial in elderly patients (≥ 70 years) affected by DLBCL defined as frail according to CGA and previously untreated.

The primary endpoint is to evaluate the efficacy of the R2 (Revlimid+Rituximab) combination in first line DLBCL patients not candidate for the standard R-CHOP (or R-CHOP like) treatments due to the frail status.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven CD20 positive Diffuse Large B-cell Lymphoma according to WHO classification (local pathologist)
2. Age ≥ 70 years
3. Previously untreated
4. CGA assessment performed before starting treatment
5. FRAIL patients defined as follows

   Age > 80 years (with UNFIT profile):

   ADL ≥ 5 residual functions and/or IADL ≥ 6 residual functions and/or CIRS: 0 comorbidity of grade 3-4 and 5-8 comorbidities of grade 2

   Age < 80 (ONLY one of the following criteria):

   ADL ≤ 4 residual functions IADL ≤ 5 residual functions CIRS: 1 comorbidity of grade 3-4 or > 8 comorbidities of grade 2
6. Ann Arbor Stage I - IV (Appendix F)
7. At least one bi-dimensionally measurable lesion defined as > 1.5 cm in its largest dimension on CT scan
8. ECOG performance status of 0- 3 (Appendix E)
9. No active hepatitis C virus (HCV) infection. In case of HCV positivity HCV-RNA is required. Only patients with HCV-RNA negative are accepted.
10. Adequate hematologic function (unless caused by bone marrow infiltrate), defined as follows:

    * Hemoglobin > 10 g/dL
    * WBC > 2500/mmc with PMN > 1000/ mmc
    * Platelets count ≥ 75000/mmc
    * Creatinine clearance ≥ 10 mL/min
11. Ability and willingness to comply with the study protocol procedure
12. Life expectancy > 6 months
13. Patients must give written informed consent.
14. Male subjects must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following investigational product discontinuation, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. Histological diagnosis different from CD20 positive Diffuse Large B-cell Lymphoma are excluded.
2. Previous exposure to cytotoxic agents
3. Suspect or clinical evidence of CNS involvement by lymphoma
4. Contraindication to the use of Rituximab or of Lenalidomide
5. HBsAg positivity; HBsAg-negative patients with anti-HBc antibody can be enrolled if Hepatitis B Virus (HBV)-DNA are negative and antiviral treatment with Lamivudine or Tenofir is provided.
6. HIV positivity
7. Active herpes zoster infection; previously infected patients is accepted only with concomitant treatment with Valacyclovir.
8. Any history of other malignancies within 5 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
9. AST /ALT > 2 x UNL; bilirubin > 2 x UNL; serum creatinine > 2.5 mg /dL
10. Creatinine clearance < 10 mL/min
11. Evidence of any severe active acute or chronic infection
12. Severe cardiac dysfunction (NYHA grade III-IV)
13. Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
14. Absence of caregivers in non-autonomous patients

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-09; Primary Completion 2020-09-22 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
ORR | 48 months
  Overall response rate (ORR) is defined as the proportion of patients with complete and partial response respectively according to Cheson 2014 (Appendix K).
  The ORR rate will be evaluated both on assessed patients and on all treated patients, considering patients without a response assessment (due to any reason) as non-responders.
  Response of R2 will be calculated for the EP according to Response Criteria for non-Hodgkin lymphoma (NHL) with CT scan; Cheson 2014; patients will be categorized into Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Non Responders (NR).
Safety: clinical relevant toxicity | 48 months
  Clinical relevant toxicity, defined as the proportion of patients experiencing a grade 3 or greater non haematological toxicity.

SECONDARY OUTCOMES:
CR | 48 months
  1) Complete response rate (CR) according to Response Criteria for non-Hodgkin lymphoma (NHL) with CT scan; Cheson 2014.
OS | 54 months
  2) Overall Survival (OS) will be defined as the time between the date of enrolment and the date of death from any cause. Patients who have not died at the time of the final analysis and patients who are lost to follow up will be censored at the date of the last contact.
PFS | 54 months
  3) Progression Free Survival (PFS) will be defined as the time between the date of enrolment and the date of disease progression, relapse or death from any cause. Responding patients, patients who are lost to follow up, who withdrawal the consent or drop-out due to adverse event will be censored at their last assessment date. Patients died due to tumor will be considered in progression. Patients died for any other cause will be censored to the death date.
  Time to event data (PFS, OS) will be estimated using the Kaplan-Meier method. The curves will be plotted and the 95% confidence interval for median time will be calculated.
EFS | 54 months
  4) Event-Free Survival (EFS), (time to treatment failure) is measured from the time from study entry to any treatment failure including disease progression, or discontinuation of treatment for any reason (eg, disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death). Responding patients, patients who are lost to follow up, who withdrawal the consent or drop-out due to adverse event will be censored at their last assessment date. Patients died due to tumor will be considered in progression. Patients died for any other cause will be censored to the death date.
Quality of life | 54 months
  5) Patients will assess their health-related quality of life (HRQoL) using two validated questionnaires: the Functional Assessment of Cancer Therapy for Lymphoma (FACT-Lym) and the Quality of life (EORTC-QLQ-C30). Items for inclusion in the lymphoma subscale were selected on the basis of symptom relevance, disease specificity, and clinical relevance.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Gini, MD, Principal Investigator — Clinica di Ematologia A.O.Universitaria Ospedali Riuniti, Ancona
Locations (18):
- Italy (18):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) - Ematologia, Meldola, Forlì-Cesena
  - A.O. C. Panico - U.O.C Ematologia e Trapianto, Tricase, Lecce
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova - IRCCS - Ematologia, Reggio Emilia, Reggio Emilia
  - Ospedale Dell'Angelo - U.O. Ematologia, Mestre, Venezia
  - Clinica di Ematologia A.O.Universitaria Ospedali Riuniti, Ancona, Ancona
  - A.O. Spedali Civili di Brescia - Ematologia, Brescia
  - IRCCS AOU S. Martino - IST - Clinica Ematologica, Genova
  - Azienda Ospedali Riuniti Papardo-Piemonte - S.C. Ematologia, Messina
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero - Universitaria Policlinico di Modena - Dipartimento di Medicina Diagnostica, Clinica e di Sanità Pubblica, Modena
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - AOU di Parma - U.O. Complessa di Ematologia, Parma
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - Ospedale delle Croci - Ematologia, Ravenna
  - Ospedale degli Infermi di Rimini - U.O. di Ematologia, Rimini
  - Policlinico Universitario Campus Bio-Medico - Area Ematologia Trapianto Cellule Staminali Medicina Trasfusionale e Terapia cellulare, Roma
  - Univ. Perugia Sede Terni - Oncoematologia, Terni
  - Ospedale ULSS 6 di Vicenza - Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gini G, Tani M, Tucci A, Marcheselli L, Cesaretti M, Bellei M, Pascarella A, Ballerini F, Petrini M, Merli F, Olivieri A, Lanza F, Annibali O, Zilioli VR, Liberati AM, Tisi MC, Arcari A, Marino D, Musuraca G, Pavone V, Fabbri A, Pozzi S, Mannina D, Plenteda C, Celli M, Luminari S. Lenalidomide plus rituximab for the initial treatment of frail older patients with DLBCL: the FIL_ReRi phase 2 study. Blood. 2023 Oct 26;142(17):1438-1447. doi: 10.1182/blood.2022019173. PMID 37418685